CLINICAL TRIAL: NCT04489927
Title: Validierung Der Messgenauigkeit Des Tcore Thermometers in Der Anwendung Nicht-invasiver Temperaturmessung gegenüber herkömmlicher Invasiver Messung Auf Der Intensivstation Bei Wachen Patienten
Brief Title: Validation of the Measurement Accuracy of the Tcore Thermometer
Acronym: T-CORE-PMCF
Status: Terminated | Type: Observational
Why Stopped: Patients couldn't be recruited (no patients with fewer available)
Sponsor: Drägerwerk AG & Co. KGaA (Industry)
Responsible Party: Sponsor
Other Study IDs: Tcore-PMCF
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tcore — Temperature Measurement of standard care versus the Tcore measurement

SUMMARY:
The aim of the study conducted at the UKSH is to investigate the measuring accuracy of the body core temperature thermometer Tcore®. Therefore the bias of the measurements to the reference measurements of the bladder catheter thermometer is determined.

DETAILED DESCRIPTION:
The aim of the study conducted at the UKSH is to investigate the measuring accuracy of the body core temperature thermometer Tcore®. Therefore the bias of the measurements to the reference measurements of the bladder catheter thermometer is determined.

Patients included are in the ICU of the UKSH and awake. They already have the reference thermometer in the catheter. The patient investigation time is limited to maximum 2 hours, SAEs will be recorded for 24 hours. The temperature of the two temperature sensors will be compared on three timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Body temperature > 34 °C
* Signed consent
* Bladder catheter with temperature sensor

Exclusion Criteria:

* Inflammation of the frontal sinus or the measuring point of the reference measurement (bladder)
* Skin irritation to the adhesive or other materials used
* medication that locally affects the body temperature or the temperature of the reference body site (barbiturates, thyroid preparations, antipsychotics, new vaccines, aspirin, acetaminophen, ibuprofen, or similar)
* Taking antipyretics in the last 120 minutes before measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in the ICU of the University Hospital Schleswig-Holstein
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Temperature | within 24 hours
  Temperature measurements with reference thermometer Tcore®

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Graf, Dr., Principal Investigator — University Schleswig-Holstein Lübeck
Locations (1):
- University Schleswig-Holstein, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No